CLINICAL TRIAL: NCT01211418
Title: Treatment of Cocaine Addiction With Integrative Meditation
Brief Title: Integrative Meditation (IM) for Cocaine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mary Bahr-Robertson, Research Supervisor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040827; R21DA025149 (NIH)
Record Dates: First submitted 2010-07-28; First posted 2010-09-29 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Cocaine Addiction
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrative Meditation (Experimental)
  Interventions: Behavioral: Integrative Meditation
- Nondirective Therapy (Active Comparator)
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: Integrative Meditation — Stage 1: Treatment Engagement and Detoxification. Use 6 breaths/minute as near resonant-frequency.
  Stage 2: Recovery and transition by reducing craving and irritability. Wk 3: introduce 16-mins IM. Wk 4: RFB & IM as a coping tool. Wk 5: add guided imagery into IM. Wk 6: review and catch-up if miss any prior sections.
  Stage 3: Revitalization and Relapse Prevention. Wk 7: customize guided imagery. Wk 8: introduce full version of IM. Wk 9: techniques of handling random thoughts during meditation and learn to separate thoughts from action. Wk 10: how to use IM techniques to handle different relapse triggers. Wk 11: different ways to integrate IM technique into daily life. Wk 12: review, feedback, and provide local sources for more meditation practice and study.
  Arms: Integrative Meditation
Behavioral: Supportive Counseling — NT is a procedure in which the therapist refrains from directing the client, but instead reflects back to the client what the latter has said. NT is chosen for this study to control for non-specific effects that show to contribute to outcome such as therapeutic alliance and therapist competency.
  The protocol for the individualized NT will mirror the layout of IM therapy -12 weekly meetings, 30 minutes each. Subjects in NT group will be instructed to do Diaphragmatic Breathing (DB) exercise and will be given assigned homework (writing journal) and track progress. DB is incorporated into the NT as treatment providing non-specific effects associated with attention and homework completion.
  Arms: Nondirective Therapy

SUMMARY:
Cocaine addiction continues to be a major problem in the U.S. with no FDA-approved pharmaceutical therapy. Finding effective treatment for cocaine addiction has long been a challenge to scientists and clinicians. Psychosocial interventions known as behavior therapies are the cornerstone of cocaine addiction treatment. However, there is an urgent need to further improve treatment outcomes, especially during early recovery and the protracted withdrawal phase of the treatment since many patients drop out or relapse during this phase. Our clinical experience and studies suggest that integrative Meditation (IM) helps reduce cravings and withdrawal symptoms and increases treatment retention. The benefit of IM is well supported by tension-reduction theory and attention-networks framework in addiction treatment. The proposed study will implement a therapy development study to add IM as a self-care component to the current outpatient treatment of cocaine addiction to improve treatment outcomes.

The specific aims of the proposed study include: 1) to conduct a 12-week controlled trial with outpatient cocaine users to assess feasibility of recruiting and retaining cocaine addicts and to determine effect size of IM-augmented treatment in comparison with Nondirective Therapy (NT) control, with both groups receiving standard outpatient treatment as usual (TAU), thereby facilitating future larger scale therapy development study; and 2) to examine the changes in attention networks and negative mood as possible mediators of treatment outcomes between the two groups.

DETAILED DESCRIPTION:
Randomization Procedure:

Subjects who meet DSM-IV cocaine dependence or abuse and other inclusion criteria will be randomly assigned to an IM or NT group, using an adaptive urn randomization procedure, which adjusts for gender, referral source (self-referred or count-mandated), psychiatric medication (yes/no), and type of cocaine addiction (polydrug vs. cocaine only). Simple randomization may not be adequate to assure a balance between the groups of known predictive indicators. While the primary basis of assignment remains randomization, urn randomization biases assignment towards balance between groups based on variables known to be related to treatment outcome when sample sizes are intermediate. Randomization reduces the possibility that one group will be assigned a disproportionate number of the few patients in certain subgroup.

Overview of the Treatment Procedure Twelve treatment sessions over 12 weeks will occur in the outpatient facility once a week, about 30 minutes each session. Treatment outcomes will be assessed at weeks 4, 8, 12, and 24 (3 months after treatment). The follow-up assessments can occur either at the outpatient facility, or at our offices in University of Maryland (Kernan Hospital). We will make the follow-up sessions at both sites equivalent to each other, and provide financial compensation for individuals who travel to our campus. For those who do not want to come to the University, we will ensure that the follow-up sessions at the treatment facility will be held in a private room separate from the location of staff and patients to ensure privacy. Subjects are clearly assured that no one at the treatment facility will have access to their treatment outcome data.

We considered having the same therapists deliver both treatments to limit therapist-specific effects independent of the actual treatment condition. Upon further consideration, we decided that this approach could potentially lead to overlap in the delivery of the two treatments and/or unintentional biases in the implementation of the control treatment. Therefore, we decided to have a total of four therapists of similar experience. Two will deliver the IM therapy, and other two will provide NT. The therapists for both groups will have similar qualifications. To prevent bias, the therapists of NT will be blinded to the study hypotheses. Treatment fidelity will be monitored through sample audio records of selected sessions to ensure the separation of treatment protocols. If diffusion occurs, further training will be utilized. To further prevent bias, none of the therapists will be involved in outcome assessment, and they will be blind to participant responses. Assessment measures will be conducted by research staff available for the study.

Description of IM Treatment Procedure Basically, IM with RFB is a combining transitions behavior therapy designed for different stages of addiction treatment. Following three stages and corresponding treatment contents will be included in the 12-week treatment.

1. Stage 1: Treatment Engagement and Detoxification (week 1-2). In our pilot study some addicts had difficult sitting still for 15-mins meditation with eyes closed, but they could do breathing exercise with eyes open. In this study we will use 6 breaths/minute as near resonant-frequency at the beginning of IM training. Each subject will receive a MP3 player with customized RFB guiding program that include waving sound (audio) and moving bar (visual) to assist the subject to do RF breathing. The subject is required to do abdominal RFB at least 15 min per day open-eye in the first week, and close-eye in the second week, then gradually switching to a combination of RFB and IM.
2. Stage 2: Recovery and transition by reducing craving and irritability (week 3-6). Based on prior feedback on RFB, from week 3 on therapist will introduce IM technique one by one to the client to practice. Week 3: introduce 16-mins IM, start with close-eye RFB, relaxing body section by section through slow breathing, and attention plus breathing to warm up lower abdomen. Week 4: RFB & IM as a coping tool, therapist helps clients find the key trigger situation for stress or relapse, and apply RFB and IM technique as a copying strategy. Week 5: add guided imagery into IM (21 mins) to help detoxify brain and body, to learn scan body part by part with increased sensation inside. Week 6: review and catch-up if miss any prior sections.
3. State 3: Revitalization and Relapse Prevention (week 7-12). Through experience of body scan by guided imagery, discuss the balance working toward change and accepting experiences that arise. Integrate IM techniques into daily life. Week 7: customize guided imagery for other problems, balance acceptance and change; Week 8: introduce full version of IM (25 mins) with technique of reversed abdominal breathing, which helps recharge the body with vital energy and calmness; conclude IM by integrating breath-mind-body into oneness - an optimal level of mind-body integration. Week 9: techniques of handling random thoughts during meditation, and learn to separate thoughts from action, a key issue in dealing with craving or relapse. Week 10: how to use IM techniques to handle different relapse triggers, do not have to act on thoughts. Week 11: different ways to integrate IM technique into daily life, make IM part of routine. Week 12: review, feedback, and provide local sources for more meditation practice and study.

The success of IM for addiction depends on therapist facilitation and quality of subject's daily practice (home-work). The description of each facilitation meeting and assigned homework are listed in the therapist manual available upon request. In general, each session the therapist will 1) get feedback from prior session and daily IM practice; 2) teach new components of IM step by step; 3) link IM technique to the addiction problem and prevention of relapse.

Nondirective Therapy (NT for control group) NT is a procedure in which the therapist refrains from directing the client, but instead reflects back to the client what the latter has said, sometimes, restating the client's remark. NT has been used as a control treatment in previous therapy development studies and was consider a good control in psychotherapy research. NT is chosen for this study to control for non-specific effects that show to contribute to outcome such as therapeutic alliance and therapist competency. Thus, both treatment conditions will contain individual therapy interaction.

The protocol for the individualized NT will mirror the layout of IM therapy -12 weekly meetings, 30 minutes each. Subjects in NT group will be instructed to do Diaphragmatic Breathing (DB) exercise and will be given assigned homework (writing journal) and track progress. DB is incorporated into the NT as treatment providing non-specific effects associated with attention and homework completion.

In short, Both IM and NT groups will get the same amount of extra contact with therapist (30 mins/week) in addition to their regular treatment, with breathing exercise (RFB or DB) and homework (IM or writing journal). Both treatment conditions will be audio-taped for evaluation of fidelity and differentiation. This design will make the study outcomes more reliable and transferable for the future therapy development studies.

ELIGIBILITY:
Inclusion Criteria:

* meets DSM-IV criteria for cocaine dependence or abuse and seeks addiction treatment
* age 18 or older
* used cocaine in the past 3 weeks, and cocaine is one of the major abused substances if using multiple drugs (urine cocaine positive at least once in the past 3 urine tests)
* is willing to adhere to the study protocol (e.g. provide urine samples, attend all visits and follow-ups in the next 6 months).

Exclusion Criteria:

* poses a current suicidal risk, including active suicidal ideation, recent suicidal behavior or suicide attempt in the past 30 days
* has a history of schizophrenia or other psychotic disorder
* unable to read or understand questions in English
* currently participates in other clinical study on addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Measurement of cocaine urine toxicology from baseline to 3 month follow-up | 3 month follow-up

SECONDARY OUTCOMES:
Compare participants' use of drugs and alcohol from baseline to 3 month follow-up | 3 month follow-up
Compare heart rate variability from baseline to 4 weeks | 4 weeks
Compare heart rate variability from 4 weeks to 8 weeks | 8 weeks
Compare heart rate variability from 8 weeks to 12 weeks | 12 weeks
Compare heart rate variability from 12 weeks to 3 month follow-up | 3 month follow-up
Change in Addiction Severity Index (ASI lite) composite scores from baseline to 3 month follow-up | 3 month follow-up
Track participant's length of time in a drug treatment program from baseline to 4 weeks | 4 weeks
Track participant's length of time in a drug treatment program from 4 weeks to 8 weeks | 8 weeks
Track participant's length of time in a drug treatment program from 8 weeks to 12 weeks | 12 weeks
Compare participants' weekly cocaine cravings from baseline to 4 weeks | 4 weeks
Compare participants' cocaine cravings from 4 weeks to 8 weeks | 8 weeks
Compare participants' cocaine cravings from 8 weeks to 12 weeks | 12 weeks
Compare participants' cocaine cravings from 12 weeks to 3 month follow-up | 3 month follow-up
Change in Beck Depression Inventory-II (BDI-II) composite scores from baseline to 4 weeks | 4 weeks
Change in Beck Depression Inventory-II (BDI-II) composite scores from 4 weeks to 8 weeks | 8 weeks
Change in Beck Depression Inventory-II (BDI-II) composite scores from 8 weeks to 12 weeks | 12 weeks
Change in Beck Depression Inventory-II (BDI-II) composite scores from 12 weeks to 3 month follow-up | 3 month follow-up
Change in participants' weekly Spielberger State-Trait Anxiety Inventory state version (STAI) composite scores from baseline to 4 weeks | 4 weeks
Change in Spielberger State-Trait Anxiety Inventory state version (STAI) composite scores from 4 weeks to 8 weeks | 8 weeks
Change in Spielberger State-Trait Anxiety Inventory state version (STAI) composite scores from 8 weeks to 12 weeks | 12 weeks
Change in Spielberger State-Trait Anxiety Inventory state version (STAI) composite scores from 12 weeks to 3 month follow-up | 3 month follow-up
Change in Self-efficacy and Self-esteem (SES) composite scores from baseline to 4 weeks | 4 weeks
Change in Self-efficacy and Self-esteem (SES) composite scores from 4 weeks to 8 weeks | 8 weeks
Change in Self-efficacy and Self-esteem (SES) composite scores from 8 weeks to 12 weeks | 12 weeks
Change in Self-efficacy and Self-esteem (SES) composite scores from 12 weeks to 3 month follow-up | 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Chen, PhD, Study Director — University of Maryland, Baltimore: Center for Integrative Medicine
Locations (3):
- United States (3):
  - Alcohol and Drug Abuse Program (ADAP), Baltimore, Maryland
  - Outpatient Addiction Treatment Service (OATS), Baltimore, Maryland
  - University of Maryland Methadone Treatment Program, Baltimore, Maryland